CLINICAL TRIAL: NCT04542278
Title: Randomized Controlled Trial of Preoperative Steroids in Autoimmune Thyroid Disease
Brief Title: Preoperative Steroids in Autoimmune Thyroid Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-0209; Protocol Ver October 2020 (Other: UW Madison); A539711 (Other: UW Madison); SMPH/SURGERY/ENDOCRINE (Other: UW Madison)
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Results first posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Thyroid Diseases
Keywords: Autoimmune disease; Graves' Disease; Hashimoto's Thyroiditis
MeSH Terms: conditions — Thyroid Diseases; Autoimmune Diseases; Graves Disease; Hashimoto Disease | interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: randomized controlled pilot study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Steroids (Active Comparator): Participants randomized to the steroid arm will be given a prescription for prednisone 20mg daily for 7 days prior to surgery, otherwise, pre-operative standard of care
  Interventions: Drug: Prednisone
- No Steroids (No Intervention): Pre-operative Standard of Care

INTERVENTIONS:
Drug: Prednisone — used to reduce inflammation
  Other Names: steroid drug
  Arms: Steroids

SUMMARY:
This pilot project will randomize a small sample of patients about to undergo surgery for their autoimmune, inflammatory thyroid disease, and determine if a short course of prednisone alters the inflammation of the gland and makes surgery less difficult. It will enroll 30 participants who will each be on study for up to 7 months.

DETAILED DESCRIPTION:
Graves' disease and Hashimoto's thyroiditis are autoimmune conditions affecting the thyroid gland. Surgery to remove the thyroid gland in these patients may be complicated by the inflammatory nature of these diseases. Prednisone is a steroid medication used to decrease inflammation of the thyroid gland in other disease states such as sub-acute thyroiditis, but has not been used systematically to reduce inflammation in patients about to undergo surgery.

This is a pilot project that proposes to randomize a small sample of patients about to undergo surgery for their autoimmune, inflammatory thyroid disease, and determine if a short course of prednisone alters the inflammation of the gland and makes surgery less difficult. This could potentially lead to better outcomes for these patients, as well as increased time to recovery and improved quality of life.

This project proposes to administer short quality of life surveys at three time points, as well as draw additional labs to measure inflammation and antibody levels at times when patients will already be getting labs drawn for clinical purposes. The purpose of this study is to generate preliminary data from which a larger, blinded, placebo-controlled trial could be designed.

These specific aims are:

* Determine the benefits and safety of preoperatively administered prednisone for patients with autoimmune thyroid disease undergoing thyroidectomy on:

  * Difficulty of surgery and rates of surgical complications
  * Serum autoantibody levels
* Longitudinally assess the impact of surgical treatment on QoL in patients with autoimmune thyroid disease

Update: Protocol amendment approved on 10-22-2020: Study team decided to omit the aim 'antibody-mediated cytokine levels' from the protocol and consent process as it became cost-prohibitive for processing and storage fees. Cytokine levels are not something typically collected or tracked in the course of clinical care, and may not be relevant. Study can proceed without this aim and will not alter the main outcome measures of antibody levels and difficulty of the operation.

ELIGIBILITY:
Inclusion Criteria:

* Graves' disease or Hashimoto's disease with positive thyroid autoantibodies (Thyroglobulin Antibody [TgAb], Thyroid peroxidase antibody [TPO], Thyroid Stimulating Ig antibody [TSI], and/or Thyrotropin Receptor antibody [TRAb]).
* Participants will be invited to join the study after the decision has been made to proceed with thyroidectomy as the clinical treatment of their autoimmune thyroid disease.

Exclusion Criteria:

* Pediatric patients < 18
* Prior treatment with radioactive iodine (RAI)
* Known diagnosis of thyroid cancer
* Diabetic patients.
* Patients on any immunosuppressive regiment (such as organ transplant patients or patients treated for other autoimmune condition)
* Pregnant patients.
* Patients being treated for active infection.
* Any patient for whom the surgeon feels steroids would provide a clear benefit (ie. Extremely high auto-antibody levels with a very large, inflamed thyroid gland) will be treated according to the clinical judgement of the surgeon. If a surgeon feels steroids are indicated and prescribes them, the patient will not be eligible for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn K Elfenbein, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Steroids | No Steroids
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Steroids | No Steroids | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (14) | 48 (15) | 44.0 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 3 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30
Number of Participants with Body Mass Index greater than or equal to 35 [Count of Participants; unit: Participants] — Body Mass Index (BMI) is a person's weight in kilograms divided by their height in meters squared. BMI over 30 is characterized as obese.
  Participants | 2 | 3 | 5
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30 (4) | 32 (10) | 31.5 (7.9)
Diagnosis [Count of Participants; unit: Participants]
  Graves' | 8 | 9 | 17
  Hashimoto's | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Thyroid Difficulty Scale Score
Description: The surgeon will fill out the "Thyroid Difficulty Scale" at the conclusion of the operation. This is a 4-item survey to rate the vascularity, friability, mobility, and glandular size of the thyroid. The total possible range of scores from 4-20, higher scores indicate increased difficulty in thyroid surgery
Time Frame: surgery occurs up to 4 weeks, data collected a conclusion of operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroids | No Steroids
Number analyzed (Participants) | 14 | 16
score on a scale | 9.8 (3.8) | 9.75 (4.0)

2. Primary Outcome: Percent Change From Baseline Mean in Autoantibody Levels
Description: Autoantibodies that may be positive include: Thyroglobulin Antibody [TgAb], Thyroid peroxidase antibody [TPO], Thyroid Stimulating Ig antibody [TSI], and/or Thyrotropin Receptor antibody [TRAb]. Any that were positive pre-op will be measured at each time point. Baseline level will be 1.
Time Frame: baseline measure day of surgery (up to 4 weeks), up to 6 weeks (2 weeks post-op), up to 10 weeks (6 weeks post-op), up to 30 weeks (6 months post-op)
Measure: Mean (Standard Deviation); unit: percent change from baseline mean
Arm/Group | Steroids | No Steroids
Number analyzed (Participants) | 14 | 16
percent change from baseline mean
  surgery to 2 weeks post op | 0.81 (0.8) | 0.78 (0.24)
  surgery to 6 weeks post-op | 0.43 (0.23) | 0.54 (0.28)
  surgery to 6 months post-op | 0.12 (0.04) | 0.24 (0.24)

3. Primary Outcome: Change in Antibody-mediated Cytokine Levels
Description: Antibody-mediated cytokine levels will be measured using a 10 cytokine panel from Luminex. Cytokines that have been implicated in other autoimmune disease include: IFN-gamma (BR29), IL-6 (BR13), IL-10 (BR22), IL-13 (BR47), IL-15 (BR63), IL-17A (BR42), and VEGF-C (BR38).
Time Frame: baseline (2-4 weeks prior to surgery), up to 4 weeks (Post Operative Day 1), up to 6 weeks (2 weeks post-op), up to 30 weeks (6 months post-op)
Population: Investigators did not collect cytokines, as originally planned, as they did not have the storage space or equipment they initially thought.
Arm/Group | Steroids | No Steroids
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Change in Short Form Health Survey (SF-12) Mental Component Score (MCS)
Description: The SF-12 is a 12-item quality of life survey to understand how the participant feels and how well they are able to do their normal activities, it is composed of the mental component score and the physical component score. Each is scored on a scale of 0-100, with higher numbers indicating higher quality of life.
Time Frame: baseline (2-4 weeks prior to surgery), up to 10 weeks (6 weeks post-op), up to 30 weeks (6 months post-op)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroids | No Steroids
Number analyzed (Participants) | 14 | 16
score on a scale
  baseline | 39.4 (11) | 35.3 (17.6)
  6 weeks post-op | 46.7 (15.7) | 38.6 (19.3)
  6 months post-op | 43.4 (16.4) | 40.3 (22.5)

5. Primary Outcome: Change in Short Form Health Survey (SF-12) Physical Component Score (PCS)
Description: as for outcome 4
Time Frame: baseline (2-4 weeks prior to surgery), up to 10 weeks (6 weeks post-op), up to 30 weeks (6 months post-op)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroids | No Steroids
Number analyzed (Participants) | 14 | 16
score on a scale
  baseline | 41.5 (10.4) | 43.2 (18.1)
  6 weeks post-op | 47.4 (14.4) | 42.7 (20.9)
  6 months post-op | 50.2 (15.8) | 44.2 (24.2)

6. Primary Outcome: Change in Thyroid-specific Quality of Life Patient-reported Outcome Measure for Benign Thyroid Disorders (ThyPRO) Score
Description: The ThyPRO survey is a quality of life measure designed to evaluate how thyroid disease has affected the participant's life. It is a 39-item survey that was scored from 0-4, higher scores indicate worse quality of life.
Time Frame: baseline (2-4 weeks prior to surgery), up to 10 weeks (6 weeks post-op), up to 30 weeks (6 months post-op)
Population: Not all participants provided survey data for all time points.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Steroids | No Steroids
Number analyzed (Participants) | 14 | 16
score on a scale
  Baseline: number analyzed (Participants) | 12 | 15
  Baseline | 2.03 [1.17 to 3.25] | 1.95 [0.67 to 2.93]
  6 weeks post-op: number analyzed (Participants) | 12 | 14
  6 weeks post-op | 1.47 [0.50 to 2.83] | 1.05 [0.36 to 2.14]
  6 months post-op: number analyzed (Participants) | 9 | 14
  6 months post-op | 1.29 [0.33 to 2.89] | 0.99 [0.21 to 2.14]

7. Secondary Outcome: Ultrasound Doppler Quantification of Blood Flow
Time Frame: baseline (2-4 weeks prior to surgery), up to 4 weeks (Post Operative Day 1)
Population: Investigators were unable to come up with a system to quantify doppler flow, so data were not collected
Arm/Group | Steroids | No Steroids
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Surgical Complications: Parathyroid Hormone (PTH) Level
Description: PTH is measured right after surgery to determine whether the nearby parathyroid glands were injured during surgery. Low PTH levels immediately after surgery are concerning for symptomatic low calcium levels, either temporarily or permanent, after thyroidectomy. Normal PTH is typically between 20-70.
Time Frame: immediately after surgery (baseline for all participants)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Steroids | No Steroids
Number analyzed (Participants) | 14 | 16
pg/mL | 52 (43) | 38 (30)

9. Secondary Outcome: Number of Participants With Surgical Complications: Recurrent Laryngeal Nerve (RLN) Injury
Time Frame: up to 4 weeks (Post Operative Day 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Steroids | No Steroids
Number analyzed (Participants) | 14 | 16
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: up to 6 months post-operatively
Arm/Group | Steroids | No Steroids
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 9/14 | 2/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Steroids (N=14) | No Steroids (N=16)
insomnia (Psychiatric disorders) | 6 | 0
mood changes (Psychiatric disorders) | 4 | 0
Gastrointestinal Upset (Gastrointestinal disorders) | 3 | 0
increased appetite (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Nerve Injury (Injury, poisoning and procedural complications) | 0 | 1
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT04542278/Prot_SAP_000.pdf